CLINICAL TRIAL: NCT00966901
Title: Assessment of Photoirritation and Photoallergic Potential of a Newly Developed Nicotine Transdermal Therapeutic System (TTS) After Single and Multiple Application and Multiple UV Exposure in Healthy Subjects. A Standard Photocontact Allergenicity Assay.
Brief Title: Photoirritation and Photoallergic Potential of a New Nicotine Patch
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Screening
Other Study IDs: A6431087; 009/05-03.NPT (Other: CRO); 2005-001641-41 (EudraCT Number)
Record Dates: First submitted 2009-08-25; First posted 2009-08-27 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Tobacco Use Cessation Devices; Radiation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Three Treatment Sites UV Exposed (Experimental): All three test sites exposed to UV radiation after patch removal. Induction: 10 J/cm2 UVA and 0.5 MED UVB, one treatment after first patch removal; and 3 MED UVB at the 5 following treatments. Challenge: 4 J/cm2 UVA and 0.5MED UVB, one treatment.( MED: Minimal Erythema Dose determined during screening)
  Interventions: Drug: Nicotine Patch; Drug: Placebo Patch; Drug: No Patch Control; Radiation: UVA and UVB irradiation

INTERVENTIONS:
Drug: Nicotine Patch — 25 mg nicotine patch applied on the assigned marked site on the lower back or buttock. Induction (23 days): six treatment applications for 24 h. Challenge (five days): one treatment application for 24 h.
  Other Names: Experimental Nicotine Patch
Drug: Placebo Patch — As a positive control, a placebo patch applied on the assigned marked site on the lower back or buttock. Induction (23 days): six treatment applications for 24 h. Challenge (five days): one treatment application for 24 h.
  Other Names: Positive Control
Drug: No Patch Control — As a negative control, a marked site on the lower back or buttock was assigned as test area, but no patch was applied.
  Other Names: Negative Control
Radiation: UVA and UVB irradiation — All three test sites exposed to UV radiation after patch removal. Induction: 10 J/cm2 UVA and 0.5 MED UVB, one treatment after first patch removal; and 3 MED UVB at the 5 following treatments. Challenge: 4 J/cm2 UVA and 0.5MED UVB, one treatment.( MED: Minimal Erythema Dose determined during screening)
  Other Names: Irradiation

SUMMARY:
An evaluation of the effects of UV exposure following the use of a new nicotine patch.

DETAILED DESCRIPTION:
An evaluation on the phototoxic potential of a newly developed nicotine patch after a single dose application followed by UV exposure, and an evaluation on the photoallergenic potential of the new nicotine patch after multiple dose applications followed by UV exposure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females between 18 and 65 years.
* Heavy smokers (more than 10 cigarettes per day) and willing to reduce the number of cigarettes smoked during the course of the study.
* Having had no febrile or infectious illness for at least seven days prior to the first administration of the investigational product.
* Women practicing one or a combination of the following methods of birth control: hormonal contraceptives, condoms, sponge, foams, jelly, diaphragm, or intrauterine device, or women who are surgically sterilized.
* Subjects having normal skin without excessive hair growth on tested areas and baseline score in skin reaction assessment of "0" on tested areas.
* Skin type I, II, or III according to Fitzpatrick.
* Evaluable MED (the lowest dose to produce mild erythema with visible borders) to UVB.
* Evidence of a personally signed and dated informed consent document indicating that the subjects have been informed of all pertinent aspects of the trial.
* Subjects who are willing to comply with scheduled visits, treatment plan and other trial procedures.

Exclusion Criteria:

* Any visible skin disorder, abnormal skin pigmentation, fissure or injury of the skin, which, in the opinion of the investigator, would interfere with the results of the trial.
* History of dermatological disease or medical conditions (in particular, any immunosuppression) which could, in the opinion of the investigator, preclude topical application of the investigational products and/or interfere with the evaluation of the test site reaction.
* History of clinically relevant psoriasis, chronic dermatitis or urticaria.
* Clinically relevant abnormal findings from the physical examination.
* Pregnant (verified by beta-HCG-test in urine) and/or nursing women.
* Any suspicion or evidence of current alcohol or drug abuse or history of alcohol or drug abuse within the last three years.
* Any current or past history of chronic or recurrent metabolic, renal, hepatic, pulmonary, gastrointestinal, neurological, endocrinological (including pheochromocytoma), immunological, psychiatric or cardiovascular disease, myopathies, epileptic seizures and bleeding tendency.
* Recent myocardial infarct (within last 3 months), unstable or deteriorating angina pectoris, coronary artery vasospasm (Prinzmetal's angina), serious cardiac arrhythmias, and acute stroke.
* History of myopathies or epileptic seizures.
* Use of any medication within four weeks prior to the first treatment or during the trial, which, in the opinion of the investigator, may influence the trial results or the safety of the subjects.
* Use of systemic or topical analgesics or antihistamines within 72 hours prior to trial enrollment (except paracetamol) or systemic or topical corticosteroids within three weeks of trial enrollment.
* Subjects having used nicotine products other than cigarettes within the three months preceding the trial.
* Participation in the treatment phase of a clinical trial within 30 days prior to the treatment phase of this trial, or within 10 times the respective elimination half-life of the investigational drug.
* Subjects who cannot avoid, throughout the duration of the trial, any swimming, any washing of the lower back (i.e., the areas which to be patched and/or irradiated during this study), usage of sauna or any intense physical activity that might result in excessive sweating.
* Any history of drug hypersensitivity, asthma, urticaria, or other severe allergic diathesis as well as current hay fever.
* Known sensitivity to adhesive tape.
* Known sensitivity to any component of the test products.
* History of irritation to topically applied products.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2005-08; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Cumulative Individual Irritation Scores after UVA and UVB exposure | 15 or 30 min, and 24, 48, and 72 hr post-application, depending on trial phase.

SECONDARY OUTCOMES:
Individual Irritation Score (IIS) | 15 min post-application, and 30 min, 24 h, 48 h, and 72 h after irradiation, depending on trial phase
Patch adhesion score | directly before patch removal
Tolerability | at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (1):
- IKP GmbH, Mannheim, Germany